CLINICAL TRIAL: NCT07062367
Title: Effect of Sevoflurane With or Without Intravenous Lidocaine Infusion Versus Propofol Anesthesia on Intracranial Pressure and Cerebral Oxygenation During Laparoscopic Hysterectomy: A Randomized Controlled Study
Brief Title: Sevoflurane With or Without Intravenous Lidocaine Infusion Versus Propofol Anesthesia on Intracranial Pressure and Cerebral Oxygenation During Laparoscopic Hysterectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Eman Ali Abd-Elsamea Elrefaey, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36265MD329/12/24
Record Dates: First submitted 2025-07-02; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Sevoflurane; Lidocaine; Propofol; Intracranial Pressure; Cerebral Oxygenation; Laparoscopic Hysterectomy
MeSH Terms: interventions — Propofol; Sevoflurane

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Propofol group (Active Comparator): Patients' anesthesia will be maintained by manually adjusted propofol infusion at a rate of 100-250 mic/kg/min for bispectral index (BIS) maintained between 40-60.
  Interventions: Drug: Propofol
- Sevoflurane plus lidocaine infusion group (Experimental): Sevoflurane with monitored anesthesia care (MAC) adjusted to maintain bispectral index (BIS) between 40-60 plus intravenous lidocaine infusion given as 2mg /kg IV bolus before induction then intraoperative infusion by a rate of 2 mg/kg/h until the end of surgery.
  Interventions: Drug: Sevoflurane plus lidocaine infusion
- Sevoflurane group (Experimental): Patients will receive sevoflurane with monitored anesthesia care (MAC) adjusted to maintain bispectral index (BIS) between 40-60.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — Patients' anesthesia will be maintained by manually adjusted propofol infusion at a rate of 100-250 mic/kg/min for bispectral index (BIS) maintained between 40-60.
  Arms: Propofol group
Drug: Sevoflurane plus lidocaine infusion — Sevoflurane with monitored anesthesia care (MAC) adjusted to maintain bispectral index (BIS) between 40-60 plus intravenous lidocaine infusion given as 2mg /kg IV bolus before induction then intraoperative infusion by a rate of 2 mg/kg/h until the end of surgery.
  Arms: Sevoflurane plus lidocaine infusion group
Drug: Sevoflurane — Patients will receive sevoflurane with monitored anesthesia care (MAC) adjusted to maintain bispectral index (BIS) between 40-60.
  Arms: Sevoflurane group

SUMMARY:
This study will be conducted to evaluate the effects of different anesthetic modalities [sevoflurane with or without intraoperative lidocaine infusion and Propofol total intravenous anesthesia (TIVA)] on intracranial pressure (ICP) and cerebral oxygenation assessed by non-invasive methods during laparoscopic hysterectomy (LH).

DETAILED DESCRIPTION:
Laparoscopic hysterectomy (LH) requires a Trendelenburg position (TP) and the creation of an artificial pneumoperitoneum (PP) by carbon dioxide insufflation.

Various studies were done to evaluate the effects of different anesthesia techniques on intracranial pressure (ICP) during LH, and most of these studies revealed that propofol total intravenous anesthesia (TIVA) was superior to inhaled anesthesia regarding reduction of ICP (ONSD).

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years.
* American Society of Anesthesiologists (ASA) physical status I and Ⅱ.
* Body mass index (BMI) ≤35.
* Females scheduled for laparoscopic hysterectomy.

Exclusion Criteria:

* Patients' refusal to participate in the study.
* Hypersensitivity and allergy to drugs of the study.
* Contraindication for optic nerve sheath diameter assessment. E.g., patient with pre-existing ophthalmic diseases, a history of ophthalmic surgery
* Any central nervous system or cardiovascular disease, severe hepatic or renal impairment
* Intraoperative circumstances, such as inability to perform optic nerve sheath diameter or conversion to open surgery
* If peak inspiratory pressure (PIP) exceeds 35.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females scheduled for laparoscopic hysterectomy
Enrollment: 90 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Optic nerve sheath diameter | After extubating the endotracheal tube (up to one hour)
  Optic nerve sheath diameter of both eyes is expressed in millimeters and will be assessed at times of: T0; baseline before induction, T1; after insertion of endotracheal tube, T2; just before pneumoperitoneum (PP), T3;30 minutes after PP and Trendelenburg position (TP),T4; 60 minutes after PP and TP,T5; Five minutes after disinflation of PP and T6;after extubating the endotracheal tube.

SECONDARY OUTCOMES:
Cerebral oxygenation | After extubating the endotracheal tube (up to one hour)
  Cerebral oxygenation of both hemispheres by near-infrared spectroscopy (NIRS). normal values 60-70% and will be assessed at times of: T0; baseline before induction, T1; after insertion of endotracheal tube, T2; just before pneumoperitoneum (PP), T3;30 minutes after PP and Trendelenburg position (TP), T4; 60 minutes after PP and TP, T5; Five minutes after disinflation of PP and T6; after extubating the endotracheal tube.
Cognitive function | 4 hours postoperatively
  Cognitive function by standardized mini mental state examination (SMMSE) preoperative, and 4hours postoperatively.
Incidence of postoperative complications | 24 hours postoperatively
  Incidence of postoperative complications such as hypotension, bradycardia, postoperative nausea and vomiting (PONV), and headache will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.